CLINICAL TRIAL: NCT01987713
Title: Chronic Conditions in Childhood Obesity Subject: An Mixed Methods Research Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 201309023
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle intervention (Experimental): the intervention strength (amount, frequency, duration) including a reduction in energy intake and an increase in physical activity level will be reported. The guidance/description of the treatment protocol, preparation and training of intervener, techniques to retain the research subjects will be covered to prevent the lack of intervention integrity. Besides, the schooler admitted in a university hospital will be invited to explore their health lifestyles and receive the intervention.
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Behavioral: lifestyle intervention — the intervention strength (amount, frequency, duration) including a reduction in energy intake and an increase in physical activity level will be reported. The guidance/description of the treatment protocol, preparation and training of intervener, techniques to retain the research subjects will be covered to prevent the lack of intervention integrity. Besides, the schooler admitted in a university hospital will be invited to explore their health lifestyles and receive the intervention.
  Other Names: amount, frequency, duration intervention

SUMMARY:
Methods: This study will be a three-year mixed methods study, including the identification of obesity issues among children with chronic conditions in the first phase study (2013/10/01-2014/07/31), development of an intervention protocol in the second phase study (2014/08/01-2015/07/31), and conduction/evaluation of an intervention of lifestyle intervention in the third phase study (2015/08/01-2016/07/31). Firstly, anthropometry, healthy lifestyles questionnaire survey on children aged 7-12 and school environment audit will be conducted. By using the literature review, meta-analysis and focus-research approaches to develop a healthy lifestyle intervention protocol in the second year program. The protocol will be tested on a sample of school-age children with asthma, to develop a school-based and family-involved healthy lifestyle intervention. Finally, the protocol will be undertaken on children with asthma aged 10-15, by using an experimental (pretest-posttest) design with repeated follow-ups. The research subjects will be randomly assign to condition of receiving intervention or control; the measurement of the outcome across 4 observations, to assess both group differences (experimental comparison), and changes within groups. The interventions consist of healthy diet (X1), regular exercise (X2), and booster energy balance-related behaviors (BEBRB) (X3). The observations start from baseline (O1), then have three observations (O2, O3, O4) at 3-month interval respectively. Outcome indicators include height, body weight, waist circumference as well as healthy life style modification present by diet record, exercise diary, healthy life environments. The research subjects will consist of randomly sampled school-age children and their fathers (or mothers), school teachers and school nurses. The approximate sample size is estimated by power analysis and dropout rate, the eligible sample size will be 200 and 160 pairs of children with their parents, school teachers and nurses in the first and third year respectively.

DETAILED DESCRIPTION:
Background: Childhood obesity is a global "public health crisis" with increasing prevalence rate in all racial, ethnic and gender groups, as well as across socioeconomic strata. Research findings indicate that over the past 30 years, the prevalence of chronic conditions in children and youths has increased. Childhood obesity impacts physical, psychological and social well-being, and also impacts the economy as well.

Purpose: The purpose of this study is to explore the healthy status, healthy lifestyles among school-age obese children of chronic conditions, then to examine the contextual factors affecting their healthy lifestyles, in order to develop a theory-informed and evidence-based intervention of school-based and family-involved intervention for obese children, and evaluate the effectiveness of interventions by using mixed methods (MM) research approach.

Methods: This study will be a three-year mixed methods study, including the identification of obesity issues among children with chronic conditions in the first phase study (2013/10/01-2014/07/31), development of an intervention protocol in the second phase study (2014/08/01-2015/07/31), and conduction/evaluation of an intervention of lifestyle intervention in the third phase study (2015/08/01-2016/07/31). Firstly, anthropometry, healthy lifestyles questionnaire survey on children aged 7-12 and school environment audit will be conducted. By using the literature review, meta-analysis and focus-research approaches to develop a healthy lifestyle intervention protocol in the second year program. The protocol will be tested on a sample of school-age children with asthma, to develop a school-based and family-involved healthy lifestyle intervention. Finally, the protocol will be undertaken on children with asthma aged 10-15, by using an experimental (pretest-posttest) design with repeated follow-ups. The research subjects will be randomly assign to condition of receiving intervention or control; the measurement of the outcome across 4 observations, to assess both group differences (experimental comparison), and changes within groups. The interventions consist of healthy diet (X1), regular exercise (X2), and booster energy balance-related behaviors (BEBRB) (X3). The observations start from baseline (O1), then have three observations (O2, O3, O4) at 3-month interval respectively. Outcome indicators include height, body weight, waist circumference as well as healthy life style modification present by diet record, exercise diary, healthy life environments. The research subjects will consist of randomly sampled school-age children and their fathers (or mothers), school teachers and school nurses. The approximate sample size is estimated by power analysis and dropout rate, the eligible sample size will be 200 and 160 pairs of children with their parents, school teachers and nurses in the first and third year respectively.

Expected outcomes: To recognize the risk factors and determinants, have an evidence-based development of school-based and family-involved lifestyle modification to better health outcomes for children with chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* 7~15years old child
* 7~15years old child's caregiver
* 7~15years old child's teacher
* 7~15years old child's nurse

Exclusion Criteria:

* not 7~15years old child
* not 7~15years old child's caregiver
* not 7~15years old child's teacher
* not 7~15years old child's nurse

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
the body weight and height to calculate the body mass index (BMI) | evaluate after intervention in 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bih-Shya Gau, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University, Taipei, Taiwan